CLINICAL TRIAL: NCT04521933
Title: Reliability of Subjective Qualitative Assessment of the Heart by Cardiac Point-of-Care Ultrasound in Comparison With Conventional Transthoracic Echocardiography
Brief Title: Reliability of Subjective Assessment of the Heart by Cardiac Point-of-Care Ultrasound
Status: Completed | Type: Observational
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Principal investigator, Masaryk Hospital Usti nad Labem
Other Study IDs: 09/2020
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Transthoracic Echocardiography
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Each participant completes a questionnaire. In the questionnaire, he performs a subjective qualitative evaluation of Point-of-Care ultrasound records of the heart.
  Each participant will complete a questionnaire in which they perform a subjective qualitative evaluation of ultrasonographic recordings of the heart.

SUMMARY:
The purpose of this study is to evaluate reliability of subjective qualitative assessment of the basic cardiac parameters by Point-pf-Care ultrasound.

DETAILED DESCRIPTION:
Subjective qualitative assessment of ventricular function, diameter of the right ventricle and the size of inferior caval vein using cardiac Point-of-Care ultrasound is commonly performed by intensivists and emergency medicine physicians during the management of the patients with shock and/or acute respiratory failure. However, very little data is available to define the reliability of this qualitative examination. The presented study aims to assess this reliability.

Physicians meeting inclusion and exclusion criteria will be sent by a questionnaire consisting of 19 ultrasound cases. Participants will be asked to perform qualitative evaluation of ultrasound findings of each case. Then, the results will be compared with quantitative measurements made by conventional transthoracic echocardiography and validity testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* physician with at least basic knowledge of cardiac Point-of-Care ultrasound who agrees to complete the questionnaire

Exclusion Criteria:

* not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians with at least basic knowledge of cardiac Point-of-Care ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Reliability of subjective qualitative assessment of the heart by Point-of-Care ultrasound in comparison with conventional transthoracic echocardiography | four weeks
  Subjective assessment of Point-of-Care ultrasound records of the heart will be performed by participants via completion of the questionnaire. Thereafter, results of the survey will be compared with the objective measurements taken by conventional transthoracic echocardiography from the same records than presented in the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk Hospital Usti nad Labem, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2015 Mar;16(3):233-70. doi: 10.1093/ehjci/jev014. PMID 25712077